CLINICAL TRIAL: NCT01482650
Title: Comparison of the Effectiveness of the BASKA Airway, a Novel Supraglottic Device, to the LMA Airway in Low Risk Female Patients
Brief Title: Comparison of the BASKA Airway, a Novel Supraglottic Device, to the LMA Airway in Low Risk Female Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, John Laffey, Professor of Anaesthesia and Critical Care, Consultant Anaesthetist, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.A. 650
Record Dates: First submitted 2011-11-25; First posted 2011-11-30 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Performance and Safety of an Airway Management Device
Keywords: Baska mask; LMA; laryngeal mask airway; supraglottic airway device

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baska mask (Experimental)
  Interventions: Device: supraglottic airway placement and use
- single use laryngeal mask airway (LMA) (Active Comparator)
  Interventions: Device: supraglottic airway placement and use

INTERVENTIONS:
Device: supraglottic airway placement and use — The investigators will place the device (Baska mask or LMA) according to a pre-defined protocol and monitor its performance intra and postoperatively.

SUMMARY:
The investigators have performed a number of studies on novel airway devices, including an observational study on the performance of a new supraglottic airway named Baska mask. In this new proposed study the investigators would like to compare directly,in a randomized clinical trial, this device with the device the investigators routinely use - the single use laryngeal mask airway - LMA, in female patients undergoing general anaesthesia.

This study will determine which device performs best, as measured by key parameters (insertion success rate, seal pressures, time to and ease of insertion, failure rate, complications etc) as regarding the performance and safety profile of the Baska mask and the LMA.

The investigators have two study hypotheses, namely (1) non-inferiority of first placement attempt success rate of Baska vs LMA; and (2) greater seal pressure of the Baska mask vs LMA.

A number of secondary endpoints will be monitored and analyzed (time to and ease of insertion, failure rate, complications etc).

DETAILED DESCRIPTION:
Airway management is essential component of the safe and efficient provision of general anaesthesia. Supraglottic airway devices have established place in the airway management.

The Baska mask is a new supraglottic airway device. It bears many of the features of the industry standard - the laryngeal mask airway (LMA), with few potential improvements:

* The cuff is not pressurized thus reducing the risk of oropharyngeal tissue damage.
* Improved cuff seal during the inspiratory phase of positive pressure ventilation which may reduce leak and make ventilation more efficient.
* An improved system for drainage of oropharyngeal contents intended to reduce the rate of lung aspiration.
* The Baska mask is inserted in neutral head position thus reducing the need for neck manipulation.
* There is integrated bite-block to reduce the risk of patients biting and blocking the airway.

The results from the observational study of the performance of the Baska mask are promising and the investigators feel a randomized comparative study against the gold standard device, the Laryngeal Mask Airway (LMA) is justified.

This study is a randomized, single blinded, controlled clinical trial. The participants will be allocated to two groups, in which the investigators will use either a single use LMA device or the Baska mask (single use).

Clinical Research Ethics Committee approval has been obtained. Suitable participants will be recruited after written informed consent and screened for inclusion and exclusion criteria.

Standard anaesthetic preassessment and anaesthesia will be provided.

Consenting patients will be randomly allocated to either of the 2 study groups.

Protocol for airway size selection and attempts at placement will be followed.

The investigators will monitor a number of parameters, including time and ease of insertion, airway seal pressure, airway leak, complications, haemodynamic and ventilatory parameters, ease of removal and other.

Follow up will be performed.

The investigators have two primary hypotheses:

1. That the BASKA mask will have an insertion success rate that is no more than 20% less than that of the single use LMA device.
2. That the seal pressure with the BASKA mask will be 40% higher than that of the single use LMA.

In addition to the above the investigators will evaluate a number of secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Written informed consent
* ASA 1-3
* No relevant allergies
* Body-mass index (BMI) 20-35
* Age 16-85
* Non-urgent surgery of planned duration 0.25-4 hrs

Exclusion Criteria:

* Inability of patient/parent to understand or consent for the trial
* Neck pathology
* Previous or anticipated problems with the upper airway or upper GI tract (reflux, hiatus hernia, oropharyngeal tumour, upper respiratory tract infection in the last 10 days)
* BMI >35
* Predicted or previously documented difficult airway
* Live Pregnancy
* Increased risk for Gastric Aspiration
* Current participation in another Clinical Study

Ages: 16 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Rate of successful placement of the supraglottic device on first attempt | Within 30minutes of commencement of general anaesthesia
  The hypothesis is that the BASKA mask will have first placement attempt success rate that is no more than 20% less than that of the single use LMA device.
Seal pressure of the supraglottic device | Within 30minutes of commencement of general anaesthesia, immediately after successful placement is accomplished.
  The investigators will measure the airway seal provided by the device used. The hypothesis is that the seal pressure with the BASKA mask will be 40% higher than that of the single use LMA.

SECONDARY OUTCOMES:
Overall rate of successful placement of the supraglottic device | Within 30minutes of commencement of general anaesthesia. Up to 3 device placement attempts are allowed.
Number of device placement attempts | Within 30minutes of commencement of general anaesthesia
User - rated Ease of insertion of the device | Within 30minutes of commencement of general anaesthesia
  the investigators will use 10cm visual analogue scale
vital parameters stability | In the period immediately before and during the first 35 minutes of the general anaesthesia
  The investigators will record noninvasive arterial oxygen saturation, heart rate and blood pressure preoperatively, after anaesthesia is induced and after the airway is placed.
Laryngeal view obtained on fiberoptic assessment | within 2hours of commencement of general anaesthesia
  The investigators will perform this where feasible.
User rated Ease of removal of the device | At the time of device removal (usually within 15 minutes before or after the end of the general anaesthesia)
  The investigators will use 10cm visual analogue scale
Complication rates | from the moment general anaesthesia commenced up to 3 days postoperatively
  Complications specifically monitored will be: blood staining, laryngospasm, lip damage, pain, dysphagia, dysphonia.
  The investigators will record other complications related to the use of the device, including but not limited to: desaturation episodes, loss of airway with need to manipulate mask/switch to alternative device, teeth damage, regurgitation, aspiration
Duration of successful insertion attepts | Within 30 minutes of commencement of general anaesthesia
  This outcome measure is defined as the period from the time device touched until successfull ventilation is achieved as per protocol.

CONTACTS AND LOCATIONS:
Overall Officials: John Laffey, FFARCSI, Principal Investigator — National University of Ireland, Galway, and Galway University Hospitals
Locations (1):
- Galway University Hospitals, Galway, Galway, Ireland